CLINICAL TRIAL: NCT05777577
Title: Immunological Profile and Microbial Markers in Evaluating the Effectiveness of Probiotic Therapy in RA Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nazarbayev University (Other)
Collaborators: Ministry of Education and Science, Republic of Kazakhstan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP14869993
Record Dates: First submitted 2023-01-31; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rheumatoid Arthritis Probiotic (RAP) (Experimental): patients with RA 30-50 yers old, who have 4 or more swollen and painful joints, who did not take probiotic and other drugs that affect the microbiome
  Interventions: Dietary Supplement: probiotic therapy
- Rheumatoid Arthritis Probiotic1 (RAP1) (Active Comparator): closest relatives (brothers and sister, children, parents) living in the same living area and corresponding to the age group, without RA, who did not take probiotic and other drugs that affect the microbiome
  Interventions: Dietary Supplement: probiotic therapy

INTERVENTIONS:
Dietary Supplement: probiotic therapy — probiotic including bifidobacterium

SUMMARY:
Rheumatoid arthritis (RA) is a common, chronic autoimmune disease that causes joint damage and deformity associated with an increased disability risk and shortened life expectancy (1). New treatment methods have significantly improved disease control, but remission is still difficult to be achieved, so new and improved treatment and diagnostic options are needed for patients stratification and prognosis. To achieve this goal, the proposed study will be aimed at studying RA main factors' relationship. The project's central theme is that microbial dysbiosis is a critical determinant of RA pathogenesis, and the interaction between human factors and the microbiome contributes to the disease risk and it's activity.

DETAILED DESCRIPTION:
The microbiome plays a fundamental role in diseases and human health. Technological advances in recent decades have expanded our understanding of microbes and their ability to form innate and acquired human immune responses. Advances in understanding the microbiome's impact on human immunity, along with the realization that inflammatory processes underlie a number of common diseases, including RA, necessitates an interdisciplinary approach to studying the interaction of humans and microbes at various levels. Modern sequencing technologies and new tools development for analyzing metagenomic data allow us to understand better the complex relationship between the dynamic microbes community inhabiting mucous tissues and the human immune system. Such analysis is especially relevant in Central Asia, since the investigators not only identified ethnic differences in risk loci, but also found that the composition of the intestinal and oral microbiota of Kazakhs is unique and significantly differs from the corresponding microbiota in other world regions, due to lifestyle factors characteristic of Kazakhstan and common to the whole Central Asia.

The main research's purpose is to study the complex relationship between microbiome dysbiosis, local and systemic inflammation in relation to RA pathogenesis and the disease activity in the Kazakhstan population. The investigators assume that patients with RA have greater dysbiosis (local microbiota violation) in the intestine and oral cavity compared to the control group, and that it is due to a greater inflammatory response and disease activity.

To consider this hypothesis, microbiome biomarkers of the oral cavity and gut in RA will be identified, RA patients immunological parameters in blood, stool and saliva samples will be analyzed, an dynamics assessment of the microbiome and immunological profile against the probiotic therapy background and an analysis of the relationships between microbiome and immunological profiles will be carried out.

The research's scientific novelty and significance consist in the study of the local and general immune status in combination with the microbiomes of the oral cavity and gut in RA. The results are likely not only to give a new insight into the relationship between human factors and pathogenic factors, but may also affect the RA diagnosis, the disease activity prognosis and inform preventive strategies. Thus, a better understanding of the complex microbial interactions with the immune system of the mucous membrane in RA can advance our understanding of RA pathophysiology, help predict future relapses, develop strategies for prevention and early diagnosis, and lead to new therapeutic directions' development aimed at the microbiome.

The results impact on the science and technology development contribute to the first comprehensive study of the RA pathogenesis in the Central Asian population. The investigators expect not only to receive important new information about the RA etiopathogenesis, but also the complex interaction that determines the pathogenesis and disease activity. The proposed study has the potential not only to improve the methods of diagnosis and monitoring of RA patients in Kazakhstan, but also can contribute to a better RA understanding in general, paving the way for personalized diagnosis and treatment of rheumatic diseases.

ELIGIBILITY:
Inclusion Criteria:

* ● age 30-50 years old

  * signed informed consent
  * Have a clinical diagnosis of RA (according to American College of Rheumatologyhttps (ACR) criteria)
  * Have been on stable RA treatment and are expected to remain on stable RA treatment during the study (ie, current medications and/or other therapies such as physical therapy are allowed, excluding immunotherapy).
  * Have at least 4 swollen and painful joints on a 64/66 scale.
  * absence of acute infectious diseases at the time of recruitment
  * absence of exacerbations of chronic diseases at the time of recruitment
  * no history of regular use of probiotic-containing products
  * no history of the use of any drugs that affect the composition of the microbiome during the last three months: antibiotics, probiotic, prebiotics, metabiotics, postbiotic

Exclusion Criteria:

* ● History of any systemic disease such as diabetes, autoimmune disease, cancer (excluding basal and squamous cell skin cancer, which have been cured) !!! taking into account the main study group

  * History of gastrointestinal or liver disease known to be associated with changes in intestinal flora
  * Use of any of the drugs listed below within the past 6 months:
* systemic antibiotics, antifungal, antiviral or antiparasitic (intravenously, intramuscularly or orally);
* oral, intravenous, intramuscular, nasal or inhaled corticosteroids;
* cytokines;
* large doses of commercial probiotic (greater than or equal to 10^8 cfu per day) - includes tablets, capsules, dragees, chewing gums or powders, where probiotic bacteria is the main component
* Use of topical antibiotics or topical steroids on the face, scalp or neck, or on the arms, forearms, hands within the previous 7 days.

  * Acute illness at the time of inclusion in the sample. Acute illness is defined as the presence of moderate or severe illness with or without fever.
  * Chronic diseases requiring current medical treatment
  * Unstable dietary history, major changes in diet during the previous month.
  * Positive test for HIV, hepatitis B virus (HBV) or hepatitis C virus (HCV).
  * Gastrointestinal surgery, excluding cholecystectomy and appendectomy in the last five years. Any major bowel resection at any time.
  * Regular urinary incontinence
  * Feeding or pregnancy.
  * Have had warts or human papillomavirus (HPV) with a confirmed diagnosis within the previous 2 years.
  * Treatment or suspected toxic shock syndrome.

Rheumatoid arthritis:

* Probable rheumatoid arthritis
* Late stage disease
* Special clinical forms of the disease: Felty's syndrome, Still's disease in adults
* Overlap syndrome, paraneoplastic syndrome

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
the oral cavity and gut microbiome | Change from Baseline the oral cavity and gut microbiome immediately after probiotic therapy
  An analysis of the biodiversity of the oral cavity and intestine will be carried out against the background of probiotic therapy: Alpha and Betta diversity according to the main indices: Chao1, Shannon, Simpson etc. The number of taxa associated with the severity of RA will be estimated using LDA. It will be analyzed to what extent probiotic therapy corrects the functional profile of the oral and intestinal microbiomes.
the oral cavity and gut microbiome | Change from Baseline the oral cavity and gut microbiome at 1 month
  An analysis of the biodiversity of the oral cavity and intestine will be carried out against the background of probiotic therapy: Alpha and Betta diversity according to the main indices: Chao1, Shannon, Simpson etc. The number of taxa associated with the severity of RA will be estimated using LDA. It will be analyzed to what extent probiotic therapy corrects the functional profile of the oral and intestinal microbiomes.

SECONDARY OUTCOMES:
the immunological profile | Change from Baseline the oral cavity and gut microbiome immediately after probiotic therapy
  the levels of the following inflammatory cytokines, chemokines and immunoglobulins will be measured in stool samples, oral swabs and blood: sCD40L (pg/mL) , EGF (pg/mL), Eotaxin/CCL11(pg/mL), FGF-2 (pg/mL), Flt-3 ligand (pg/mL), Fractalkine (pg/mL), G-CSF (pg/mL), GM-CSF (pg/mL), GRO (pg/mL), IFN-α2 (pg/mL), IFN-γ (pg/mL), IL-1α (pg/mL), IL-1β (pg/mL), IL-1ra (pg/mL), IL-2 (pg/mL), IL-3 (pg/mL), IL-4 (pg/mL), IL-5 (pg/mL), IL-6 (pg/mL), IL-7(pg/mL), IL-8(pg/mL), IL-9(pg/mL), IL-10(pg/mL), IL-12 (p40)(pg/mL), IL-12 (p70)(pg/mL), IL-13(pg/mL), IL-15(pg/mL), IL-17A(pg/mL), IP-10(pg/mL), MCP-1(pg/mL), MCP-3(pg/mL), MDC (CCL22)(pg/mL), MIP-1α(pg/mL), MIP-1β(pg/mL), PDGF-AA(pg/mL), PDGF-AB/BB(pg/mL), RANTES(pg/mL), TGF-α(pg/mL), TNF-α(pg/mL), TNF-β(pg/mL), VEGF(pg/mL), IgA (g/L), IgG1-G4 (g/L), IgM (g/L).
the immunological profile | Change from Baseline the oral cavity and gut microbiome at 1 month
  the levels of the following inflammatory cytokines, chemokines and immunoglobulins will be measured in stool samples, oral swabs and blood: sCD40L (pg/mL) , EGF (pg/mL), Eotaxin/CCL11(pg/mL), FGF-2 (pg/mL), Flt-3 ligand (pg/mL), Fractalkine (pg/mL), G-CSF (pg/mL), GM-CSF (pg/mL), GRO (pg/mL), IFN-α2 (pg/mL), IFN-γ (pg/mL), IL-1α (pg/mL), IL-1β (pg/mL), IL-1ra (pg/mL), IL-2 (pg/mL), IL-3 (pg/mL), IL-4 (pg/mL), IL-5 (pg/mL), IL-6 (pg/mL), IL-7(pg/mL), IL-8(pg/mL), IL-9(pg/mL), IL-10(pg/mL), IL-12 (p40)(pg/mL), IL-12 (p70)(pg/mL), IL-13(pg/mL), IL-15(pg/mL), IL-17A(pg/mL), IP-10(pg/mL), MCP-1(pg/mL), MCP-3(pg/mL), MDC (CCL22)(pg/mL), MIP-1α(pg/mL), MIP-1β(pg/mL), PDGF-AA(pg/mL), PDGF-AB/BB(pg/mL), RANTES(pg/mL), TGF-α(pg/mL), TNF-α(pg/mL), TNF-β(pg/mL), VEGF(pg/mL), IgA (g/L), IgG1-G4 (g/L), IgM (g/L).

IPD SHARING:
Plan to Share IPD: No